Official Title: A brief intervention targeting anhedonia in adolescents: a feasibility randomised controlled trial

NCT ID: not yet assigned

**Document: Consent Forms** 

Document Date: 20/05/2022

## **CONSENT FORM FOR PARTICIPANTS IN RESEARCH STUDIES**



Please complete this form after you have read the Information Sheet and/or listened to an explanation about the research.

This consent form is for participants A new psychological programme to improve mood and build self-esteem: stage 1 King's College Research Ethics Committee Ref: HR-19/20-14899

Thank you for considering taking part in this research. The person organising the research must explain the project to you before you agree to take part. If you have any questions arising from the Information Sheet or explanation already given to you, please ask the researcher before you decide whether to join in. You will be given a copy of this Consent Form to keep and refer to at any time.

Please tick or initial I confirm that I understand that by ticking/initialling each box I am consenting to take part in this element of the study. I understand that it will be assumed that unticked/initialled boxes mean that I DO NOT consent to take part in that part of the study. I understand that by not giving consent for any one element, I may not be able to take part in the study. Please tick or initial 1. \* I agree that I have read the information sheet about the study and am happy with the answers to my questions. 2. \*I understand that taking part is voluntary and I am free to stop at any time without giving a reason. I also understand that I can withdraw my data until 31st June 2022. 3. \*I consent to the processing of my personal information for the purposes explained to me. I understand that my information will be handled in accordance with the terms of the UK Data Protection Act 1998. 4. \*I understand that certain members of the researcher's university may look at my information. I understand that my answers are private and will not be shared with anyone else unless the researcher is concerned about me. I understand that it will not be possible to identify me in any scientific articles. 5. \*I understand that my responses are confidential unless I mention something that concerns the project researcher of my safety or the safety of someone else, they are obliged to break confidentiality and inform my parents and/or relevant school teachers. 6. \*I understand that I must not take part if I meet any of the criteria that have been detailed in the information sheet and explained to me by the researcher. 7. \*I consent to my school being informed about my participation I am invited to take part in Stage 2 8. \*I consent to being contacted by email or phone if I am invited to the next stage of the project. (Please give your details for which you prefer to be contacted on)

Email address:

Mobile number:

| Full Name of Participant | Date | Signature |
|--------------------------|----------|-----------|
| Full Name of Researcher | <br>Date | Signature |

## **CONSENT FORM FOR PARTICIPANTS IN RESEARCH STUDIES**

Please complete this form after you have read the Information Sheet and/or listened to an explanation about the research.



This consent form is for participants

A new psychological programme to improve mood and build self-esteem: stage 2 King's College Research Ethics Committee Ref: HR-19/20-14899

Thank you for considering taking part in this research. The person organising the research must explain the project to you before you agree to take part. If you have any questions arising from the Information Sheet or explanation already given to you, please ask the researcher before you decide whether to join in. You will be given a copy of this Consent Form to keep and refer to at any time.

Please tick or initial I confirm that I understand that by ticking/initialling each box I am consenting to take part in this element of the study. I understand that it will be assumed that unticked/initialled boxes mean that I DO NOT consent to take part in that part of the study. I understand that by not giving consent for any one element, I may not be able to take part in the study. Please tick or initial 1. \* I agree that I have read the information sheet about the study and am happy with the answers to my questions. 2. \*I understand that taking part is voluntary and I am free to stop at any time without giving a reason. I also understand that I can withdraw my data until 31st June 2022. 3. \*I consent to the processing of my personal information for the purposes explained to me. I understand that my information will be handled in accordance with the terms of the UK Data Protection Act 1998. 4. \*I understand that certain members of the researcher's university may look at my information. I understand that my answers are private and will not be shared with anyone else unless the researcher is concerned about me. I understand that it will not be possible to identify me in any scientific articles. 5. I agree that King's College London researchers can contact me in the future to take part in other similar research (optional). 6. I consent to my answers in the assessments being audio recorded (optional). 7. I consent to my sessions being audio recorded (optional). 8. I consent to the audio recordings being used for the purposes of teaching and training other professionals (optional). 9. \*I consent to being contacted by email or phone if I am invited to the next stage of the project. (Please give your details for which you prefer to be contacted on) Email address: or Mobile number: 10. \*I understand that my responses are confidential unless I mention something that concerns the project researcher of my safety or the safety of someone else, they are obliged to break confidentiality and inform my parents and/or relevant school teachers. 11. \*I understand that I must not take part if I meet any of the criteria that have been detailed in the information sheet and explained to me by the researcher.

| Full Name of Participant | Date Date | Signature |
|--------------------------|-----------|-----------|
| Full Name of Researcher | <br>Date | Signature |

## **CONSENT FORM FOR PARENTS/GUARDIANS IN RESEARCH STUDIES**



This form is for parents/guardians.

Please complete these forms after you have read the Information Sheets and/or listened to an explanation about the research. If you provide your consent on the Stage 2 consent form and your child is eligible to take part in the programme, we will invite your child to take part and will contact you to make you aware of this.

A new psychological programme to improve mood and build self-esteem: stage 1 King's College Research Ethics Committee Ref: HR-19/20-14899

Thank you for considering for your child to take part in this research. The person organising the research must explain the project to you before you agree for your child to take part. If you have any questions arising from the Information Sheet or explanation already given to you, please ask the researcher before you decide whether to let your child join in, their contact details are on the information sheet. You will be given a copy of this Consent Form to keep and refer to at any time.

Please tick or initial

I confirm that I understand that by ticking/initialling each box I am consenting to my child taking part in this element of the study. I understand that it will be assumed that unticked/initialled boxes mean that I DO NOT consent to my child taking part in that part of the study. I understand that by not giving consent for any one Please tick element, my child may not be able to take part in the study. or initial 12. \* I agree that I have read the information sheet about the study and am happy with the answers to my questions. 1. \*I understand that my child's participation is voluntary and they are free to stop at any time without giving a reason. I also understand that my child can withdraw their data until 31st June 2023. 13. \*I consent to the processing of my child's personal information for the purposes explained to me. I understand that my child's information will be handled in accordance with the terms of the UK Data Protection Act 1998. 14. \*I understand that certain members of the researcher's university may look at my child's information. I understand that my child's answers are private and will not be shared with anyone else unless the researcher is concerned about my child. I understand that it will not be possible to identify my child in any scientific articles. 15. I agree that King's College London researchers can contact me (if my child is still under 16) and my child in the future to take part in other similar research (optional). 16. I consent to my child's answers in the assessments being audio recorded (this will apply if your child is invited to Stage 2) (optional). 17. I consent to my child's sessions being audio recorded (this will apply if your child is invited to Stage 2) (optional). 18. I consent to the audio recordings being used for the purposes of teaching and training other professionals (this will apply if your child is invited to Stage 2) (optional)

| the project researcher of their confidentiality and inform mys | 19. *I understand that my child's responses are confidential unless they mention something that concerns the project researcher of their safety or the safety of someone else, the researcher is obliged to break confidentiality and inform myself as the parent/guardian and/or relevant school teachers (this will apply if your child is invited to Stage 2). | |
|---|---|---|
| • | · | neet any of the criteria that have been detailed searcher (this will apply if your child is invited to |
| Full Name of parent/guardian | <br>Date | <br>Signature |
| Full Name of Researcher Date | <br>e | Signature |